CLINICAL TRIAL: NCT01232946
Title: Cooperation of Insulin and GLP-1 on Myocardial Glucose Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Kieren Mather, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1105005578
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Myocardial metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Liraglutide; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Iiraglutide (Experimental): Type 2 diabetic subjects will be assigned to 3 months of treatment with 1.8mg liraglutide administered once daily in addition to background metformin 2000mg/day. PET measurements of myocardial glucose uptake will take place at the end of treatment.
  Interventions: Drug: liraglutide
- insulin detemir (Experimental): Type 2 diabetic subjects will be assigned to 3 months of treatment with insulin detemir administered twice daily in addition to background metformin 2000mg/day. PET measurements of myocardial glucose uptake will take place at the end of treatment.
  Interventions: Drug: insulin detemir
- Liraglutide plus insulin detemir (Experimental): Type 2 diabetic subjects will be assigned to 3 months of treatment with a combination of liraglutide and insulin detemir in addition to background metformin 2000mg/day. PET measurements of myocardial glucose uptake will take place at the end of treatment.
  Interventions: Drug: liraglutide plus insulin detemir

INTERVENTIONS:
Drug: liraglutide — 1.8mg subcutaneous qd for 3 months
  Other Names: Victoza
  Arms: Iiraglutide
Drug: insulin detemir — 5units subcutaneous bid titrated to fasting glucose of <130mg/dL for 3 months
  Other Names: Levemir
  Arms: insulin detemir
Drug: liraglutide plus insulin detemir — liraglutide 1.8mg subq qd plus insulin detemir 5units bid titrated to fasting blood glucose <130mg/dL for 3 months.
  Other Names: Vyctoza plus Levemir
  Arms: Liraglutide plus insulin detemir

SUMMARY:
27 Type 2 diabetic subjects (HbA1c 7.5 - 9.5%) currently treated with diet and exercise alone or with oral antidiabetic agents will be randomly assigned to one of three treatment groups: insulin detemir, liraglutide, or liraglutide plus detemir (9 subjects per group), on a background of metformin 2000 mg per day. After 3 months' treatment, PET measurements of myocardial fuel selection will take place, under fasting conditions in the morning following that day's treatment injection(s).

DETAILED DESCRIPTION:
The investigators will test the hypothesis that effects of liraglutide plus insulin detemir on myocardial fuel selection will be greater than the effects of either agent alone. 27 Type 2 diabetic subjects (HbA1c 7.5 - 9.5%) currently treated with diet and exercise alone or with oral antidiabetic agents will be randomly assigned to one of three treatment groups: insulin detemir, liraglutide, or liraglutide plus detemir (9 subjects per group). All subjects will undergo an initial standardization of background treatment to metformin 2000 mg per day, followed by randomized assignment to 3 months' treatment with liraglutide 1.8 mg/day (once daily each morning, tapering up according to label instructions) and/or detemir (administered twice daily, initially at 10 units per day then titrated to achieve fasting morning glucose readings below 130 mg/dL). PET measurements of myocardial fuel selection will take place at the end of this treatment period, under fasting conditions in the morning following that day's treatment injection(s).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic
* 18-50 years
* BMI > 25kg/m2
* HbA1c 7.0-10.0%
* Treated with up to 2 oral agents

Exclusion Criteria:

* Chronic illness or infection (other than diabetes mellitus)
* Known coronary artery disease, structural heart disease or abnormal ECG on screen.
* Treatment with >2 antihypertensive agents or blood pressure >140/95 on two occasions during screening
* History of claustrophobia, musculoskeletal or other factors which would result in an inability to comfortably remain within the PET scanner gantry for the duration of the imaging protocol.
* Occupational, investigational or other known radiation exposure which together with the planned radiologic studies, will result in greater than 500 mrem total exposure in a 12 month period.
* Current pregnancy
* Treatment with GLP-1 agonist or DPP4 inhibitor within the past 6 months
* Known intolerance to GLP-1 agonist
* Personal history of pancreatitis, personal or family history of medullary thyroid carcinoma, or other contraindications to liraglutide treatment.
* Recognized microvascular complications (neuropathy, nephropathy, retinopathy).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieren J Mather, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana Clinical Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mather KJ, Considine RV, Hamilton L, Patel NA, Mathias C, Territo W, Goodwill AG, Tune JD, Green MA, Hutchins GD. Combination GLP-1 and Insulin Treatment Fails to Alter Myocardial Fuel Selection vs. Insulin Alone in Type 2 Diabetes. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3456-3465. doi: 10.1210/jc.2018-00712. PMID 30020461

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iiraglutide | Insulin Detemir | Liraglutide Plus Insulin Detemir
Started | 9 | 10 | 11
Completed | 9 | 9 (1 participant died unrelated to study) | 9 (2 withdrew after baseline measurements)
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iiraglutide | Insulin Detemir | Liraglutide Plus Insulin Detemir | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (5.3) | 52.1 (8.6) | 49.2 (9.0) | 51.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 8 | 17
  Male | 7 | 2 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 7 | 13
  White | 6 | 6 | 2 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 27
HbA1c, % [Mean (Standard Deviation); unit: %] | 7.59 (0.96) | 7.00 (0.79) | 8.13 (0.99) | 7.57 (0.91)

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Glucose Uptake
Description: PET measurements of myocardial glucose uptake will be done after 3 months of exposure to liraglutide, insulin detemir, or liraglutide plus insulin detemir
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: umol/g/min
Arm/Group | Iiraglutide | Insulin Detemir | Liraglutide Plus Insulin Detemir
Number analyzed (Participants) | 9 | 9 | 9
umol/g/min | 0.055 [0.0186 to 0.1047] | 0.0399 [0.0129 to 0.0494] | 0.0373 [0.0085 to 0.0455]
Statistical Analysis 1: Comparison: Iiraglutide vs Insulin Detemir vs Liraglutide Plus Insulin Detemir; Test type: Superiority; p = 0.65, Kruskal-Wallis

2. Primary Outcome: Myocardial Fatty Acid Oxidation Rate
Description: as for outcome 1
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: umol/g/min
Arm/Group | Iiraglutide | Insulin Detemir | Liraglutide Plus Insulin Detemir
Number analyzed (Participants) | 9 | 9 | 9
umol/g/min | 0.1019 [0.0803 to 0.1399] | 0.1234 [0.0711 to 0.1836] | 0.0992 [0.0801 to 0.1352]
Statistical Analysis 1: Comparison: Iiraglutide vs Insulin Detemir vs Liraglutide Plus Insulin Detemir; Test type: Superiority; p = 0.065, Kruskal-Wallis

3. Primary Outcome: Myocardial Fatty Acid Esterification Rate
Description: as for outcome 1
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: umol/g/min
Arm/Group | Iiraglutide | Insulin Detemir | Liraglutide Plus Insulin Detemir
Number analyzed (Participants) | 9 | 9 | 9
umol/g/min | 0.00274 [0.00236 to 0.01234] | 0.00358 [0.00249 to 0.00917] | 0.00146 [0.00038 to 0.00863]
Statistical Analysis 1: Comparison: Iiraglutide vs Insulin Detemir vs Liraglutide Plus Insulin Detemir; Test type: Superiority; p = 0.80, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Study interval is ~4 months for each participant. Total study duration from first participant entered to last participant completed was ~3 yrs.
Arm/Group | Iiraglutide | Insulin Detemir | Liraglutide Plus Insulin Detemir
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iiraglutide (N=9) | Insulin Detemir (N=10) | Liraglutide Plus Insulin Detemir (N=11)
Gastrointestinal intolerance (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iiraglutide (N=9) | Insulin Detemir (N=10) | Liraglutide Plus Insulin Detemir (N=11)
Gastrointestinal intolerance (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-10-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT01232946/Prot_SAP_000.pdf